CLINICAL TRIAL: NCT06674590
Title: Effects of Motor Relearning Program Versus Proprioceptive Neuromuscular Facilitation on Balance and Gait in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/49
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Chronic Stroke; Proprioceptive Neuromuscular Facilitation; Balance; Gait; Gait Speed
Keywords: Stroke; Motor relearning program; Proprioceptive neuromuscular facilitation; balance; gait; gait speed; stride length; cadence; cycle time
MeSH Terms: conditions — Stroke | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group A (Experimental): It includes participants receiving proprioceptive neuromuscular facilitation physical therapy for chronic stroke patient's for balance and gait parameter for a period of 6 weeks.
  Interventions: Procedure: Proprioceptive Neuromuscular Facilitation
- Experimental group B (Experimental): It includes participants receiving motor relearning program physical therapy for chronic stroke patient's for balance and gait parameter for a period of 6 weeks.
  Interventions: Procedure: Motor Relearning Program

INTERVENTIONS:
Procedure: Proprioceptive Neuromuscular Facilitation — PNF of 30 minutes duration will given in a single session. Pelvic anterior elevation and posterior depression of the hemiplegic side. rhythmic initiation slow reversal agonistic reversals Pelvic anterior depression and posterior elevation of the hemiplegic side. The first diagonal (D1): Flexion and extension The second diagonal (D2): Flexion and extension 4 session per week
  Arms: Experimental group A
Procedure: Motor Relearning Program — Motor Relearning Programme (MRP) This is a task-oriented approach to help the control of movement, focusing on the relearning of daily activities.
  Arms: Experimental group B

SUMMARY:
A randomized control trial will be done on diagnosed stroke patients of chronic stage in DHQ Hospital Mirpur and FF Hospital Rawalpindi physical therapy Department.The purpose of the study is to determine Effects of Motor Relearning Program Versus Proprioceptive Neuromuscular Facilitation on Balance and Gait in Stroke .

Subjects will complete Berg Balance Scale (BBS). 10-meter walk test for gait speed will be used for measuring walking speed in meters per second over a short distance, Timed-Up-And-Go (TUG) Test will be used for test of functional mobility and gait parameter. All these measures will be taken at baseline, then after 6 weeks of intervention. There will be 4 sessions per week. The control group will receive Group Motor relearning programe while the Study Group (B) will receive Proprioceptive Neuromuscular Facilitation(PNF)

DETAILED DESCRIPTION:
OBJECTIVES:

The objectives of this study are:

1. To determine the effects of Motor Relearning program Versus Proprioceptive Neuromuscular Facilitation for Improving Balance in stroke patient.
2. To determine the effects of Motor Relearning program Versus ProprioceptiveNeuromuscular Facilitation on Gait Parameters in stroke patient.

HYPOTHESIS:

Alternate hypothesis:

Motor Relearning program as compared to Proprioceptive Neuromuscular Facilitation effective for balance and gait parameter in chronic stroke patient.

Null hypothesis:

Motor Relearning program as compared to Proprioceptive Neuromuscular Facilitation not effective for balance and gait parameter in chronic stroke patient.

Research Design: Experimental study. Randomized Control Trial

Clinical setting: DHQ Hospital Mirpur , Fauji Foundation Hospital . Study duration: 1 year

Selection Criteria:

Inclusion Criteria

1. more than 6 month post stroke
2. Can ambulate 25 feet/10 meter (with or without assistive device).
3. Age between 25 to 65 years.
4. Grades for MAS (Grade 2 0r less )/stage of brunstrom approach (stage 4 or up )

Exclusion Criteria

1. History of neurologic disease other than the chronic stroke.
2. Orthopedic disorder involving any joint of lower limbs that interfere with study.
3. Gross visuospatial deficits .
4. Unhealed fracture of lowerlimb .
5. Peripheral arterial occlusive disease.
6. Uncontrolled hypertension and diabetes .

Sampling technique: Non Proability Purposive sampling

Outcome Measures:

Data will be collected on Demographics and general information Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function .

10-meter walk test for gait speed The 10 Meter Walk Test is a performance measure used to assess walking speed in meters per second over a short distance.

Timed-Up-And-Go (TUG) Test:

test of functional mobility in which the participant stands up from a standard armchair, walks to a line on the floor 3 m away, turns around, walks back to the chair, and sits dow

Control group (A) = MRP divided into different task , duration will be 30 minutes. MRP for sitting to standing MRP for stand to sit MRP for walking Training of hip extension throughout stance phase Training of knee control for stance phase Training of lateral horizontal pelvic shift Training of flexion of knee at start of swing phase Training of knee extension and foot dorsiflexion at heel strike Practice of walking Transference of training into daily Experimental Group (B) =PNF of 30 minutes duration will given in a single session.

Pelvic anterior elevation and posterior depression of the hemiplegic side. rhythmic initiation slow reversal agonistic reversals Pelvic anterior depression and posterior elevation of the hemiplegic side. The first diagonal (D1): Flexion and extension The second diagonal (D2): Flexion and extension

Data analysis techniques:

The data will be analyzed through SPSS 21 and Data would be analyzed based on the study design chosen that is random control experimental study.

A printed questionnaire will be provided to the participents after obtaining written consent and providing adequate explanation regarding the study, after which the data will be presented in the form of graphs or tables.

Significance of the study:

Proprioceptive Neuromuscular Facilitation compared to motor relearning program for chronic stroke patient may prove effectiveness in term of balance and gait parameters.

This study will help the practitioner to use the best treatment options for treating patients with stroke problem.

The results of the study will add to the literature about the effect of Proprioceptive Neuromuscular Facilitation as compared to motor relearning program for of balance and gait parameter in stroke patient.

ELIGIBILITY:
Inclusion Criteria:

* more than 6 month post stroke
* both male and female
* Can ambulate 25 feet/10 meter (with or without assistive device).
* Age between 25 to 65 years.
* Grades for MAS (Grade 2 0r less )/stage of brunstrom approach (stage 4 or up )

Exclusion Criteria:

* History of neurologic disease other than the chronic stroke.
* Orthopedic disorder involving any joint of lower limbs that interfere with study.
* Gross visuospatial deficits .
* Unhealed fracture of lowerlimb .
* Peripheral arterial occlusive disease.
* Uncontrolled hypertension and diabetes

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
gait parameter | 6 weeks
  measurements of how a person walks, by using 10 meter walk test and TUG

SECONDARY OUTCOMES:
Balance | 6 weeks
  an even distribution of weight enabling someone or something to remain upright and steady by using BBS

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan